CLINICAL TRIAL: NCT07375550
Title: Adherence Determinants of Medication Non-Adherence Among Patients With Chronic Diseases at Community Pharmacy Settings in Egypt: A Multicenter Cross-Sectional Study
Brief Title: Determinants of Medication Non-Adherence Among Patients With Chronic Diseases in Egyptian Community Pharmacies
Acronym: ADHER-EG
Status: Not yet recruiting | Type: Observational
Sponsor: Egyptian Chinese University (Other)
Responsible Party: Principal Investigator, Sarah Sabry Hashem Nafea, Principal Investigator: Assisstant Professor of Pharmacy Practice Faculty of pharmacy and Drug Technology, Egyptian Chinese University
Other Study IDs: 3
Record Dates: First submitted 2025-12-30; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-12

CONDITIONS: Chronic Disease
Keywords: Chronic Disease; Egypt; Community pharmacy; Medication Adherence
MeSH Terms: conditions — Chronic Disease; Medication Adherence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Medication non-adherence among patients with chronic diseases is a major public health concern and is associated with poor disease control, increased complications, and higher healthcare costs. Community pharmacists play an important role in supporting patients' medication use through counseling and education; however, the determinants of medication non-adherence among patients attending community pharmacies in Egypt are not well characterized.

This multicenter, cross-sectional study aims to assess the prevalence of medication non-adherence and identify factors associated with non-adherence among adult Egyptian patients with chronic diseases attending community pharmacy settings. Medication adherence will be evaluated using the Adherence in Chronic Diseases Scale (ACDS), along with sociodemographic, clinical, and medication-related factors. The findings are expected to provide evidence to inform strategies for improving medication adherence and optimizing chronic disease management in community pharmacy practice in Egypt.

DETAILED DESCRIPTION:
Chronic diseases represent a substantial burden on healthcare systems and require long-term pharmacological treatment to prevent complications and maintain optimal health outcomes. Effective management of these conditions relies heavily on patients' adherence to prescribed medication regimens. Medication non-adherence is common worldwide and is associated with disease progression, increased hospitalizations, reduced quality of life, and increased healthcare costs.

Community pharmacists are accessible healthcare professionals who are well positioned to support medication adherence through patient education, counseling, and follow-up. Despite this, medication non-adherence remains prevalent, and the factors contributing to non-adherence among patients with chronic diseases in Egypt have not been adequately studied. Sociodemographic characteristics, clinical factors, medication-related issues such as adverse effects, and the availability and quality of pharmacist counseling may all influence adherence behavior.

This study is designed as a multicenter, cross-sectional investigation conducted in community pharmacies across major Egyptian cities, including Cairo, Alexandria, and Giza. The study population includes adult patients aged 18 to 80 years who have been diagnosed with at least one chronic disease and are currently receiving pharmacological treatment for their condition.

Data will be collected using a structured, interviewer-administered questionnaire. Information gathered will include sociodemographic characteristics, clinical and medication history, and exposure to medication counseling. Medication adherence will be assessed using the Adherence in Chronic Diseases Scale (ACDS), a validated tool for evaluating adherence behaviors in patients with chronic conditions.

The primary outcome of the study is the prevalence of medication non-adherence among patients with chronic diseases attending community pharmacies. Secondary outcomes include identification of factors associated with medication non-adherence, such as medication side effects, patient-related characteristics, and pharmacist-provided counseling. Data analysis will be performed using SPSS software, with binary logistic regression applied to identify significant predictors of medication adherence. Statistical significance will be set at a p-value of less than 0.05.

The study is observational and poses minimal risk to participants. Ethical approval will be obtained from the relevant local ethics committee, and the study will be conducted in accordance with applicable ethical guidelines. Written informed consent will be obtained from all participants prior to enrollment. Participant confidentiality will be maintained through anonymization of collected data.

The results of this study are expected to generate important local evidence on medication adherence among Egyptian patients with chronic diseases and to support the development of targeted interventions and policies aimed at enhancing medication adherence and improving health outcomes in community pharmacy settings.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 80 years.
* Diagnosed with at least one chronic disease requiring long-term pharmacological treatment.
* Currently receiving at least one prescribed medication for a chronic condition.
* Attending a participating community pharmacy during the study period.
* Able and willing to provide written informed consent.

Exclusion Criteria:

* Patients with cognitive impairment or mental conditions that limit their ability to understand the study procedures or complete the questionnaire.
* Patients who refuse or are unable to provide written informed consent.
* Patients who are acutely ill and unable to participate at the time of data collection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 to 80 years who have been diagnosed with at least one chronic disease and are receiving long-term pharmacological treatment. Participants will be recruited from community pharmacy settings across multiple Egyptian cities Eligible patients are those attending participating community pharmacies during the study period and who are capable of understanding the study procedures and providing written informed consent. The study population reflects a real-world sample of patients managing chronic conditions in community pharmacy practice in Egypt.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Medication Non-Adherence Among Patients with Chronic Diseases | Through study completion, an average of 1 month (cross-sectional assessment)
  Medication non-adherence will be assessed using the Adherence in Chronic Diseases Scale (ACDS), a validated questionnaire designed to evaluate patients' adherence behaviors toward prescribed medications for chronic conditions. The outcome will be expressed as the proportion of participants classified as non-adherent and adherent based on ACDS scoring, and analyzed in relation to sociodemographic and clinical factors.

SECONDARY OUTCOMES:
Determinants and Predictors of Medication Non-Adherence in Patients with Chronic Diseases | Through study completion, an average of 1 month (cross-sectional assessment)
  analysis will be used to identify significant predictors of medication non-adherence as measured by the Adherence in Chronic Diseases Scale (ACDS).

IPD SHARING:
Plan to Share IPD: No